CLINICAL TRIAL: NCT04070313
Title: A Phase II Study of S-1 Adjuvant Chemotherapy in Patients With Resected Pancreatic Cancer in Taiwan
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study treatment is to use TS-1 (mono-chemotherapy agent) in adjuvant setting for pancreatic cancer, which may be less clinical benefit compared to combination therapy according to current trend at investigators' discretion.
Sponsor: TTY Biopharm (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTYTG1709
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Resected Pancreatic Cancer; Pancreatic Cancer; Adjuvant Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S-1 (Experimental): single-arm
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — Eligible patients will receive S-1 orally 80-120 mg/day (depending on patient's body surface area (BSA)) on day 1 to 28 in a 6-week cycle.

SUMMARY:
To verify the efficacy of S-1 adjuvant chemotherapy in resectable pancreatic cancer.

* Primary Endpoint: Relapse-free survival (RFS)
* Secondary Endpoints: 2-year survival rate, 2-year relapse-free survival (RFS) rate, safety profile

ELIGIBILITY:
Inclusion Criteria:

1. Patients with resected adenocarcinoma pancreatic cancer that was histologically verified.
2. Patients with macroscopic total resection of the primary tumor, and confirmed local residual tumor classified as R0/R1.
3. Absence of distant metastases and malignant ascites
4. Adequate oral intake
5. Age of 20 years or above
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or1
7. Adequate hematopoietic which is defined as below,

   * White blood cell count: 3,000/mm3, ≤ 12,000/mm3
   * Platelet count: 100,000/mm3
   * Hemoglobin: 8.0 g/dL
   * ANC: 1500/mm3
8. CA19-9 ≤ 100 U/mL
9. Absence used of chemotherapy or radiotherapy
10. Within 10 weeks following resection of pancreatic cancer
11. Written informed consent given

Exclusion Criteria:

1. Patient previously received adjuvant therapy for pancreatic cancer
2. Patient previously received S-1 treatment and concurrent using other fluoropyrimidine-group anti-cancer drugs, combination therapies with them (such as folinate plus Tegafur-Uracil combination therapy)
3. Recurrence prior to registration
4. Moderate or more severe pleural effusion or ascites upon abdominal CT
5. Inadequate hepatic function which is defined as below:

   * Total bilirubin greater than 1.5 times the ULN
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)greater than 2.5 times the ULN
6. Inadequate renal function which is defined as below:

   Creatinine clearance rate (CCr) < 60 mL/min
7. Heart failure of Class III (Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea.) or Class IV (Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.) according to the New York Heart Association functional classification
8. Other serious complications such as active peptic ulcer, paresis of intestine or any others
9. Pulmonary fibrosis or interstitial pneumonia clearly observed
10. Uncontrolled watery diarrhea Whether a patient has diarrhea 4 or more times a day while receiving adequate supportive therapy will be used as the indicator to determine whether watery diarrhea is inadequately controlled.
11. Blood transfusion within 2 weeks prior to registration
12. Myocardial infarction within 6 months following documentation of pancreatic cancer
13. An active infectious disease (pyrexia of 38°C or higher, etc.), including active Hepatitis B or C.

    * Active HBV: HBeAg positive or HBeAg negative but HBV DNA > 2000 IU/mL.
    * Active HCV: Anti-HCV Ab positive
14. Poorly controlled diabetes mellitus:

    Fasting blood sugar ≥ 200 mg/dL or HbA1c ≥ 10.0 %
15. Participation in the study by the patient is judged difficult due to a complicating psychiatric disorder or psychological symptoms
16. Patient is using drainage.
17. Serious drug allergy or hypersensitivity to the ingredients of S-1
18. Other malignancy with the exception of non-melanoma skin cancer or cervical carcinoma in situ within 5 years prior to registration
19. Pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential. Fertile women of childbearing potential unless using a reliable and appropriate contraceptive method throughout the treatment period and for three months following cessation of treatment.
20. Man who is willing to conceive a child during the treatment period.
21. On flucytosine, phenytoin or warfarin potassium treatment.
22. Participation in another clinical trial with any investigational drug within 30 days prior to registration.
23. Patients who were judged to be ineligible as the subjects of this study by the investigators

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | 2 years
  The time from registration to the time of initial detection of relapse or death from any causewhichever came first, assessed up to 2 years

SECONDARY OUTCOMES:
2-year survival rate | 2 years
  The number of patient who occur relapse or death from any cause, whichever comes first before end of 2 years
2-year relapse-free survival (RFS) rate | 2 years
  the percentage of people in a study who are alive 2 years after their diagnosis or the start of treatment
safety profile | 2 years
  The incidence and percentage of patients with at least one occurrence of preferred term will be included,according to the most severe NCI-CTCAE v5.0 grade

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Chang Gung Memorial Hospital_Linkou, Linkou District
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taiwan, Taipei